CLINICAL TRIAL: NCT04486300
Title: Seasonal Variations and Different Treatment Protocols OF Intussusception In Children: Our Center Experience.
Brief Title: Seasonal Variations and Different Treatment Protocols OF Intussusception In Children:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Ahmed ElSayed A. Moustafa, Associate Professor of Pediatric Surgery, Minia University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 100500323
Record Dates: First submitted 2020-06-28; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Intussusception
Keywords: Intussusception, Pediatric surgery, Pneumoreduction
MeSH Terms: conditions — Intussusception | interventions — Laparotomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Season of presentation (No Intervention): Comparison of number of presented cases in each season
- Intervention (Active Comparator): Surgical intervention of failed Pneumatic cases is done
  Interventions: Procedure: Pneumatic reduction and Laparotomy

INTERVENTIONS:
Procedure: Pneumatic reduction and Laparotomy — Pneumatic reduction is the main intervention for suitable cases and If failed a laparotomy exploration and surgical reduction is done to save life
  Arms: Intervention

SUMMARY:
Background: Intussusception remains a common cause of bowel obstruction in children and results in significant morbidity and mortality if not promptly treated. There is a paucity of prospective studies regarding childhood intussusception. This study describes the seasonal variation and management outcomes of childhood intussusception.

METHODS: This was A prospective study of all patients admitted and treated for childhood intussusception aged < 12 year intussusception from January 2014 to December 2018 was conducted in El-Minia University Pediatric surgery unit. Data about the ages of the patients, sex, clinical presentation, duration of symptoms before presentation, mode of treatment, outcome of treatment, and incidence of recurrence were recorded and analyzed.

DETAILED DESCRIPTION:
A prospective study from January 2014 to December 2018 was conducted in 470 cases in El-Minia University Pediatric surgery unit. All pediatric patients (up to 14 years old) hospitalized with diagnosis of bowel intussusception were included in the study. The clinical records included: age, gender, signs, symptoms, and number of any previous episodes of intussusception and their treatment, concomitant pathologies and intolerance, ultrasound data, laboratory parameters and performed treatment.

An ultrasonography was performed when patients presented suspicion symptoms and signs of intussusception, in order to confirm the diagnosis and exclude other causes. Diagnosis was based on the presence of the "target sign" on vertical section on ultrasound images. Collected data included location and diameter of the intussusception, free fluid in abdomen and presence of visible pathological lead point. If diagnosis was confirmed, the management and treatment depended on the patients' situation, in patients complaining of severe dehydration, high grade fever and other signs of septicemia the conservative treatment was contraindicated and direct surgical treatment was performed. For children in good general conditions initial Pneumatic reduction under continuous imaging monitoring using a C-arm device was attempted; if reduction failed or unstable vital signs were observed, enema was discontinued and surgical management was proposed. If intussusception recurrence was observed in the next hours, Pneumatic reduction was performed again whenever possible.

Treatment After fluid and electrolyte correction, Pneumatic reduction was performed by using air through an 18 F urinary catheter applied to the rectum under continuous imaging guidance by C-arm. With child in a supine position, a Foley catheter was introduced in the rectum and maintained by inflating its balloon with 40 ml saline; the buttocks were joined with a band aid in order to avoid leaks. The rectal cannula was connected to Sphygmomanometer inflatable cuff initially about 80 mmHg increasing up to a maximum of 120. The passage of air into the ileum through the ileocecal valve ensures successful reduction. No time limit was imposed on the duration of the procedure; however, cessation of retrograde movement of the intussusception for more than 15 minutes was regarded as a failed attempt. The procedure was repeated 20 minutes later, with a maximum of 3 attempts.

All children were kept under medical supervision, no oral intake was permitted for the following 24 hours and intravenously fluids and antibiotics were given. After 12 to 24 hours ultrasonography was repeated to exclude early recurrence.

ELIGIBILITY:
Inclusion Criteria:

* All patients in the pediatric age group (<14 years).
* Proved diagnosis of acute intussusception.
* Completion of patient's data in the medical records.

Exclusion Criteria:

* Other concomitant disease.
* Refused cases

Ages: 18 Months to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 470 (Actual)
Dates: Start 2014-01-14 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2020-03-07 (Actual)

PRIMARY OUTCOMES:
Time of presentation | 2 years
  Seasons with high presented cases

SECONDARY OUTCOMES:
Surgery | 2 Years
  If we needed Invasive Intervention or Classic reduction

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: data will be available for 10 years
Access Criteria: open Access Journal